CLINICAL TRIAL: NCT02870023
Title: How Does Strength Training and Balance Training Affect Gait Function and Fatigue in Patients With Multiple Sclerosis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: VIA University College (Other); TrygFonden, Denmark (Industry); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 14695664
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Balance training (Experimental): All sessions will start with a ten minute warm-up on either a treadmill or a cycle.
  The balance intervention will be conducted in stations/domains where balance is challenged in the five different functions: standing, walking, sit to stand, stepping, and a station that exercises vestibular and gaze control.
  Progression is achieved by adding exercises with increased balance requirements and by adding additional motoric and cognitive tasks to the exercises-dual-tasking.
  Intensity of the exercises is defined from an error-rate where an adequate level is 20-40 percent.
  The intervention is conducted according to a standardized framework that describes examples of exercises and progressions.
  Interventions: Other: Balance training
- Strength training (Experimental): All sessions will start with a ten minute warm-up on a stationary bicycle, followed by strength training of primary muscle synergies in the lower extremities. All exercises will be performed on machines with patients sitting or lying, adequately supported. The exercises are leg press, knee extension, hip flexion, hamstring curl, and hip extension. Exercises are performed with a fast concentric phase and a slow eccentric phase..
  Set, repetition, and load:
  * Weeks 1 and 2, 3 sets of 10 repetitions at a load of 15 repetitions maximum (RM)
  * Weeks 3 and 4, 3 sets of 12 repetitions at a load of 12RM
  * Weeks 5 and 6, 4 sets of 12 repetitions at a load of 12RM
  * Weeks 7 and 8, 4 sets of 10 repetitions at a load of 10RM
  * Weeks 9 and 10, 4 sets of 8 repetitions at a load of 8RM.
  Interventions: Other: Strength training
- Control group (No Intervention): On a waitlist. After ten weeks of waiting, and intervention that contains 50 percent strength training and 50 percent balance training begins.

INTERVENTIONS:
Other: Balance training
  Arms: Balance training
Other: Strength training
  Arms: Strength training

SUMMARY:
Introduction: Multiple sclerosis (MS) is characterized by decreased strength and motor control, and compromised gait function. Reduced walking speed, balance, and fatigue are the cardinal symptoms. In rehabilitation, strength and balance training are commonly used. There is increasing scientific support of strength training for improving walking function. The evidence for balance training remains flawed. It is known that neurological damage in MS leads to increased cognitive processing in the planning of movements, which predisposes fatigue. Since fatigue is also associated with impaired balance, it can be hypothesized that motoric/balance training with an emphasis on cognitive load can affect gait and fatigue.

Purpose: The aim of the study is to determine whether there is a differentiated effect between strength and balance training measured by motor function, strength, balance, and fatigue.

DETAILED DESCRIPTION:
People with MS experience a wide variety of symptoms including impaired muscle strength and balance, fatigue, impaired cognition, depression and spasticity. Of these, impaired balance and severe fatigue are described as two of the most debilitating symptoms leading to limitations in activities such as upright posture and gait. Generally, pharmacological symptomatic treatment has not proven efficient in the treatment of balance problems, fatigue and walking impairments, with the exception that Fampridine has beneficial effects on gait performance in a subgroup of patients. Consequently, non-pharmacological interventions that effectively target these symptoms are warranted.

In the last decade progressive resistance training (PRT) has proven to be one of the promising interventions in patients with MS showing a consistent and positive effect on muscle strength. However, the effect of PRT on functional outcomes are heterogeneous but with promising effects on daily activities such as walking and chair rise. The evidence for a beneficial effect of PRT on balance and postural control is divergent and yet inadequately investigated. Regarding fatigue, a recent Cochrane review reported that one could expect improvements in MS fatigue after exercise interventions, despite methodological flaws in the existing literature, but only few studies evaluating PRT were located.

Another promising intervention is task specific training of motor function that is widely used by physiotherapists in neurorehabilitation. In this study protocol, motor function is limited to gait related functions with a particular focus put on balance and motor control, why the term Balance and Motor Control Training (BMCT) is applied. There is no universally accepted definition of human balance, but balance defined as "the inherent ability of a person to maintain, achieve or restore a specific state of balance and not to fall, with reference to the motor and sensory systems and to the physical properties of the person", is applied in this study.

Effects obtained from BMCT partly result from plastic changes in the nervous system. To induce such effects, repetition of a simple task only has limited efficiency in order to improve performance. Once a task has been learned to a certain level, further practice of the same task will not be accompanied by further induction of plasticity and little is therefore gained by continued practice of the task. To provide challenges that ensures continued learning, training exercises have to progress from simple movement trajectories to more complex movements, that also incorporates goal setting. Moreover, it has been shown that shaping and variation of tasks in combination with feedback on movement quality is of great importance for the learning outcome. The underlying concept for performing BMCT is, therefore, that improved motor control will optimize the movement strategy, which further leads to improved gait function.

Regarding the effects of BMCT on fatigue, there are diverging results in the literature, but the literature on BMCT for patients with MS is generally of low quality with an inadequate description of interventions, why further studies are warranted.

Interestingly, the principles of task specific training do fundamentally contrast the principles of PRT, that normally consist of monotonous movement patterns performed under heavy loading for a low number of repetitions. Consequently, studies comparing the effects of BMCT and PRT on gait function would add to the current literature as no studies doing so could be located. Such a comparison would help clarify whether potential effects are overlapping or differentiated and would therefore help guiding future rehabilitation interventions in persons with MS.

The primary objective of this study is, therefore, to investigate and compare the effects of 10 weeks of PRT to BMCT on gait function, balance and fatigue in mobility limited persons with MS.

It is hypothesized that PRT will be superior in improving maximal straight gait speed, whereas BMCT will have a greater impact on balance, fatigue, and more complex walking tasks that include elements of balance and coordination.

ELIGIBILITY:
Inclusion criteria

* Diagnosed with multiple sclerosis.
* Expanded Disability Status Scale (EDSS) 2.0-6.5 and min. 2.0 in the functional system "pyramidal function".
* Able to walk 100 m.
* Able to manage own transportation in relation to weekly training and tests.
* Six spot step test score > 8 sec. or Timed 25 foot walk > 5 sec.

Exclusion criteria

* Co-morbidity in terms of dementia and alcohol abuse.
* Attack within the last eight weeks.
* Systematic intensive rehabilitation/training within the last three months.
* Adjustment of medication within two months before inclusion. This applies only for medication that affects gait performance and spasticity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in gait speed measured by "Six Spot Step Test" | At baseline and again after 10 weeks
  Six Spot Step Test
Change in gait speed measured by "Timed 25 Foot Walk" | At baseline and again after 10 weeks
  Timed 25 Foot Walk

SECONDARY OUTCOMES:
Fatigue | At baseline and after 10 weeks
  Fatigue: Fatigue is measured according to the Danish version of the modified fatigue impact scale.
Endurance | At baseline and after 10 weeks
  Six-minute walk
Self-evaluated gait function | At baseline and after 10 weeks
  MS walking scale
Temporospatial measures | At baseline and after 10 weeks
  Gait in fastest and self-selected speed is recorded by a Qualisys system for 3D analysis. Determinants are step and stride length, step width, time in swing and stance, gait speed, and hip and knee angles during gait.
Balance - static | At baseline and after 10 weeks
  (modified) Clinical test for sensory interaction and balance (CTSIB). The test is conducted on a force plate that measures movement of center of pressure (COP). Outcome is length of COP trajectory and elliptic area.
Balance - functional | At baseline and after 10 weeks
  Mini BESTest
Balance - confidence | At baseline and after 10 weeks
  The Activities-specific Balance Confidence Scale
Strength | At baseline and after 10 weeks
  Maximum voluntary isometric contraction in knee flexion and extension. Maximum voluntary isometric and isokinetic contraction in dorsal and plantar flexion.

OTHER OUTCOMES:
General health | At baseline and after 10 weeks
  Short-Form Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Callesen, PT, MHSc, Principal Investigator — University of Aarhus
Locations (1):
- Department of Public Health - Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boes MK, Sosnoff JJ, Socie MJ, Sandroff BM, Pula JH, Motl RW. Postural control in multiple sclerosis: effects of disability status and dual task. J Neurol Sci. 2012 Apr 15;315(1-2):44-8. doi: 10.1016/j.jns.2011.12.006. Epub 2012 Jan 10. PMID 22236888
- [Background] Claros-Salinas D, Dittmer N, Neumann M, Sehle A, Spiteri S, Willmes K, Schoenfeld MA, Dettmers C. Induction of cognitive fatigue in MS patients through cognitive and physical load. Neuropsychol Rehabil. 2013;23(2):182-201. doi: 10.1080/09602011.2012.726925. Epub 2012 Nov 16. PMID 23153337
- [Background] Penner IK, Bechtel N, Raselli C, Stocklin M, Opwis K, Kappos L, Calabrese P. Fatigue in multiple sclerosis: relation to depression, physical impairment, personality and action control. Mult Scler. 2007 Nov;13(9):1161-7. doi: 10.1177/1352458507079267. PMID 17967844
- [Background] Andreasen AK, Stenager E, Dalgas U. The effect of exercise therapy on fatigue in multiple sclerosis. Mult Scler. 2011 Sep;17(9):1041-54. doi: 10.1177/1352458511401120. Epub 2011 Apr 5. PMID 21467189
- [Background] Corporaal SH, Gensicke H, Kuhle J, Kappos L, Allum JH, Yaldizli O. Balance control in multiple sclerosis: correlations of trunk sway during stance and gait tests with disease severity. Gait Posture. 2013 Jan;37(1):55-60. doi: 10.1016/j.gaitpost.2012.05.025. Epub 2012 Aug 5. PMID 22874664
- [Background] Kelleher KJ, Spence W, Solomonidis S, Apatsidis D. The characterisation of gait patterns of people with multiple sclerosis. Disabil Rehabil. 2010;32(15):1242-50. doi: 10.3109/09638280903464497. PMID 20156050
- [Background] Hebert JR, Corboy JR. The association between multiple sclerosis-related fatigue and balance as a function of central sensory integration. Gait Posture. 2013 May;38(1):37-42. doi: 10.1016/j.gaitpost.2012.10.015. Epub 2012 Nov 28. PMID 23200463
- [Background] Motl RW, Pilutti LA. The benefits of exercise training in multiple sclerosis. Nat Rev Neurol. 2012 Sep;8(9):487-97. doi: 10.1038/nrneurol.2012.136. Epub 2012 Jul 24. PMID 22825702
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Huisinga JM, Filipi ML, Stergiou N. Supervised resistance training results in changes in postural control in patients with multiple sclerosis. Motor Control. 2012 Jan;16(1):50-63. doi: 10.1123/mcj.16.1.50. PMID 22402220
- [Background] Cattaneo D, Jonsdottir J, Zocchi M, Regola A. Effects of balance exercises on people with multiple sclerosis: a pilot study. Clin Rehabil. 2007 Sep;21(9):771-81. doi: 10.1177/0269215507077602. PMID 17875557
- [Background] Paltamaa J, Sjogren T, Peurala SH, Heinonen A. Effects of physiotherapy interventions on balance in multiple sclerosis: a systematic review and meta-analysis of randomized controlled trials. J Rehabil Med. 2012 Oct;44(10):811-23. doi: 10.2340/16501977-1047. PMID 22990349
- [Derived] Callesen J, Cattaneo D, Brincks J, Dalgas U. How does strength training and balance training affect gait and fatigue in patients with Multiple Sclerosis? A study protocol of a randomized controlled trial. NeuroRehabilitation. 2018;42(2):131-142. doi: 10.3233/NRE-172238. PMID 29562556